CLINICAL TRIAL: NCT01407328
Title: The Effect of the Shoulder Arthroscopic Surgery on Respiratory Mechanics
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gwak Mi Sook, Professor, Samsung Medical Center
Other Study IDs: 2011-06-031
Record Dates: First submitted 2011-07-05; First posted 2011-08-02 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Shoulder Arthroscopic Surgery
Keywords: shoulder arthroscopic surgery; respiratory discomfort; airway obstruction; restrictive pathology; diaphragm palsy
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
During shoulder arthroscopic surgery, extravasation of irrigation fluid can occur around the shoulder and trachea, compressing the upper airway. Although the extravasation is generally reabsorbed asymptomatically within 12 hours, there are cases that lead to reintubation or life-threatening complications. Furthermore, the soft tissue edema around the shoulder may extend to the thoracic cage, compress the chest and induce the respiratory distress immediately after surgery. The investigators attempt to determine the effect of shoulder arthroscopic surgery on respiratory mechanics. Changes in respiratory mechanics and arterial blood gases were measured and compared before and after the shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
Currently, most shoulder surgeries are performed with arthroscopy. The advantages of shoulder arthroscopic surgery are decreased blood loss due to minimal incision for scope, a reduced operation time, minimization of surgical stress, and rapid recovery time after surgery. During shoulder arthroscopic surgery, extravasation of irrigation fluid can occur around the shoulder and trachea, compressing the upper airway. Although the extravasation is generally reabsorbed asymptomatically within 12 hours, there are cases that lead to reintubation or life-threatening complications. Furthermore, the soft tissue edema around the shoulder may extend to the thoracic cage, compress the chest and induce the respiratory distress immediately after surgery. From these facts, the mechanism of respiratory discomfort after shoulder arthroscopic surgery may be because the upper airway obstruction or restrictive pathology due to direct compression of thoracic cage by the soft tissue edema. There have been no studies on the respiratory effect of shoulder arthroscopic surgery. We have observed frequent and severe respiratory discomfort after the shoulder arthroscopic surgery. Therefore, in this study we attempt to determine the effect of shoulder arthroscopic surgery on respiratory mechanics. Changes in respiratory mechanics and arterial blood gases were measured and compared before and after the shoulder arthroscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic shoulder rotator cuff repair surgery
* American society of anesthesiologist (ASA) class I or II
* Patients under 70 yrs.

Exclusion Criteria:

* Patients older than 70 yrs,
* Patients with anatomical derangement of upper airway,
* Patients with pulmonary or cardiac disease,
* Patients with a history of laryngeal or tracheal surgery or hemodynamic instability

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing arthroscopic shoulder rotator cuff repair surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Static compliance | before and after arthroscopic surgery, an expected average of 80 minutes
  Static compliance (mL/cmH2O) before and after the arthroscopic surgery
  ,Static compliance = tidal volume delivered / (plateau pressure - PEEP)
dynamic compliance | before and after arthroscopic surgery, an expected average of 80 minutes
  dynamic compliance (mL/cm H2O) before and after the arthroscpic surgery
  ,dynamic compliance = tidal volume delivered / (peak pressure - PEEP)

SECONDARY OUTCOMES:
inspiratory tidal volume | before and after arthroscopic surgery, an expected average of 80 minutes
  inspiratory tidal volume (ml) before and after the arthroscpic surgery
expiratory tidal volume | before and after arthroscopic surgery, an expected average of 80 minutes
  expiratory tidal volume (ml) before and after the arthroscpic surgery
peak inspiratory pressure | before and after arthroscopic surgery, an expected average of 80 minutes
  peak inspiratory pressure (cm H2O) before and after the arthroscpic surgery
physiologic dead space | before and after arthroscopic surgery, an expected average of 80 minutes
  physiologic dead space (VD/VT) before and after arthroscopic surgery
  ,VD/VT = (PaCO2 - PeCO2)/PaCO2, PeCO2 = mixed expired CO2
plateau airway pressure | before and after arthroscopic surgery, an expected average of 80 minutes
  plateau airway pressure (cmH2O) before and after arthroscopic surgery
Mean airway pressure | before and after arthroscopic surgery, an expected average of 80 minutes
  Mean airway pressure (cm H2O) before and after arthroscopic surgery
positive end expiratory pressure | before and after arthroscopic surgery, an expected average of 80 minutes
  positive end expiratory pressure (cmH2O) before and after arthroscopic surgery
inspiratory resistance | before and after arthroscopic surgery, an expected average of 80 minutes
  inspiratory resistance (cmH2O/L sec) before and after arthroscopic surgery
expiratory resistance | before and after arthroscopic surgery, an expected average of 80 minutes
  expiratory resistance (cmH2O/ L sec)before and after arthroscopic surgery
peak inspiratory flow | before and after arthroscopic surgery, an expected average of 80 minutes
  peak inspiratory flow (L/min) before and after arthroscopic surgery
peak expiratory flow | before and after arthroscopic surgery, an expected average of 80 minutes
  peak expiratory flow (L/min) before and after arthroscopic surgery
Work of breathing | before and after arthroscopic surgery, an expected average of 80 minutes
  Work of breathing (J/L) before and after arthroscopic surgery
end tidal CO2 | before and after arthroscopic surgery, an expected average of 80 minutes
  end tidal CO2 (mmHg) before and after arthroscopic surgery
arterial oxygen tension | before and after arthroscopic surgery, an expected average of 80 minutes
  arterial oxygen tension (mmHg) measured by arterial blood gas analysis
arterial CO2 tension | before and after arthroscopic surgery, an expected average of 80 minutes
  arterial CO2 tension (mmHg)as measured by arterial blood gas analysis
forced vital capacity (FVC) | before and after general anesthesia, an expected average of 120 minutes
  forced vital capacity measured by portable spirometry
forced expiratory volume for 1 second (FEV1) | before and after general anesthesia, an expected average of 120 minutes
  forced expiratory volume for 1 second (FEV1)measure by portable spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Mi Sook Gwak, M.D.,Ph.D., Principal Investigator — Samsung Medical Center; Won Ho Kim, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea